CLINICAL TRIAL: NCT05029271
Title: InPen User Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP338
Record Dates: First submitted 2021-08-11; First posted 2021-08-31 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Type 1
Keywords: Multiple Daily injections; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Single Arm exploratory and descriptive study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- InPen with Guardian 4 System Arm (Other): All subjects will move from phase 1 to phase 4 of the study.
  Phase 1:
  Blinded Continuous Glucose Monitoring (CGM) will be utilized while subjects are on their current MDI therapy.
  Phase 2:
  All subjects will utilize a smart bolus insulin pen injector (InPen™) and app with dose calculator (InPen™ Diabetes Management App).
  Phase 3:
  Subjects will continue on the InPen and InPen App utilizing the HCP insights gained during the titration follow-up visit.
  Phase 4:
  All subjects will utilize the InPen™ with the Guardian™ 4 system.
  Interventions: Device: InPen with Guardian 4 System

INTERVENTIONS:
Device: InPen with Guardian 4 System — Subjects will receive the InPen™ and InPen™ Diabetes Management App combined with the Guardian™ 4 system.

SUMMARY:
The purpose of this study is to evaluate the user experience of InPen™ with InPen™ Diabetes Management App and Guardian 4 system in adult patients with type 1 diabetes for the design of a future pivotal study.

DETAILED DESCRIPTION:
This study is a multi-center, single arm study in insulin-requiring adult subjects with type 1 diabetes treated with MDI (basal and bolus) therapy.

The total study duration will be approximately 10 weeks long for each participant.

The study consists of a run-in (phase 1) and study phases 2, 3 and 4.

Phase 1:

The purpose of the run-in phase is to collect baseline HbA1c and blinded Continuous Glucose Monitoring (CGM) data while subjects are on their current MDI therapy.

Phase 2:

All subjects will utilize a smart bolus insulin pen injector (InPen™) and app with dose calculator (InPen™ Diabetes Management App), and will continue their own SMBG, iscCGM or RT-CGM for two weeks.

Phase 3:

Subjects will continue on the InPen and InPen App for another two weeks utilizing the HCP insights gained during the titration follow-up visit.

Phase 4:

All subjects will utilize the InPen™ system consisting of:

* InPen™ and InPen™ Diabetes Management App
* Guardian™ 4 system (RT-CGM)
* Guardian™ 4 sensor
* Guardian™ 4 transmitter
* Guardian™ 4 app

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18-75 years at time of screening
2. Subject is on MDI therapy (defined as ≥ 3 insulin injections per day and on a basal/bolus regimen) ≥1 year prior to screening
3. Subject has a clinical diagnosis of type 1 diabetes for 1 year prior to screening
4. Subject has a Glycosylated hemoglobin (HbA1c) less than 10% as assessed by local lab <15 days prior to screening or at time of screening visit
5. Subject is on MDI therapy with

   1. SMBG,
   2. Continuous Glucose Monitoring (CGM), or
   3. Intermittent Scanning CGM (iscCGM)
6. Subject is willing to upload data from a BG meter, must have internet access and a compatible computer system that meets the requirements for uploading data at home.
7. Subject is willing and able to sign and date informed consent, comply with all study procedures, and wear all study devices, as required during the study.
8. Subject is willing to take or switch to one of the following insulins:

   1. Humalog™* (insulin lispro injection)
   2. NovoLog™* (insulin aspart)

Exclusion Criteria:

1. Women of child-bearing potential who have a positive pregnancy test at screening or plan to become pregnant during the course of the study.
2. Women who are breastfeeding.
3. Subject has any unresolved adverse skin conditions in the area of sensor placement (e.g. psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
4. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or device in the last 2 weeks before enrollment into this study, as per investigator judgment.
5. Subject is currently abusing illicit drugs, marijuana, alcohol or prescription drugs (other than nicotine), per investigator judgment.
6. Subject has any other disease or condition that may preclude the patient from participating in the study, per investigator judgment.
7. Subject is legally incompetent, illiterate or vulnerable person.
8. Research staff involved with executing the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Endpoints are exploratory and descriptive related to time in glycemic range. | Above endpoints will be categorized by daytime and night-time and overall (24hour).
  Percentage of Time spent within range with sensor glucose (SG) between 70-180 mg/dL (3.9-10.0 mmol/L)

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Örebro University Hospital, Örebro
  - NU-Hospital Group, Uddevalla
  - Frolunda specialist hospital, Västra Frölunda

IPD SHARING:
Plan to Share IPD: No